CLINICAL TRIAL: NCT01247389
Title: Incisional Hernia After Midline Versus Transverse Extraction Incision in Laparoscopic Colectomy: A Pilot Randomized Trial
Brief Title: Incisional Hernia After Midline Versus Transverse Extraction Incision in Laparoscopic Colectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Dr. Liane S. Feldman, MD, McGill University Health Centre/Research Institute of the McGill University Health Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10-183-SDR
Record Dates: First submitted 2010-11-23; First posted 2010-11-24 (Estimated); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Laparoscopic Colectomy
Keywords: laparoscopy; colon resection; incisional hernia
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- midline incision (Active Comparator)
  Interventions: Procedure: laparoscopic colectomy
- transverse incision (Active Comparator)
  Interventions: Procedure: laparoscopic colectomy

INTERVENTIONS:
Procedure: laparoscopic colectomy — Laparoscopic segmental colectomy with planned abdominal extraction site

SUMMARY:
Incisional hernia (IH) is a common complication of midline laparotomy. Despite the hope that laparoscopic colon resection would result in fewer incisional hernias, prospective studies demonstrate a similar incidence to open surgery. Observational studies suggest that the rate of incisional hernia after laparoscopic colon resection may be reduced with the use of a transverse compared to a midline extraction incision. However, no randomized trails are available, and a midline extraction incision for hemicolectomy remains the standard current approach. The investigators hypothesize that the use of a lower abdominal transverse muscle splitting incision for specimen extraction in laparoscopic colon surgery will result in fewer incisional hernias compared to a midline periumbilical extraction incision.

ELIGIBILITY:
Inclusion Criteria:

* scheduled laparoscopic partial colectomy where an abdominal extraction incision is planned

Exclusion Criteria:

* previous laparotomy
* rectal resection or anastamosis
* planned pfannenstiel extraction incision
* single site surgery
* planned or performed stoma
* BMI >35 kg/m2
* ASA 4-5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 165 (Actual)
Dates: Start 2011-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incisional hernia | one year

SECONDARY OUTCOMES:
surgical site infection | one month
body image | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Montreal General Hospital, Montreal, Quebec, Canada